CLINICAL TRIAL: NCT03376204
Title: Characteristics of Underlying Pain Mechanisms in Patients With Bronchiectasis: a Cross-sectional Study
Brief Title: Pain Mechanisms in Patients With Bronchiectasis
Status: Withdrawn | Type: Observational
Why Stopped: It has been impossible to recruit any participants fulfilling both the inclusion criteria. Therefore, the current study protocol is no longer valid.
Sponsor: Universidad San Jorge (Other)
Responsible Party: Principal Investigator, Víctor Doménech, Physiotherapy Lecturer at San Jorge University and Researcher at iPhysio Research Group from San Jorge University., Universidad San Jorge
Other Study IDs: PI17/0290
Record Dates: First submitted 2017-10-19; First posted 2017-12-18 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Bronchiectasis; Respiratory Disease
Keywords: Bronchiectasis; Pain mechanisms; Pressure pain threshold; Referred pain
MeSH Terms: conditions — Bronchiectasis; Respiration Disorders; Pain, Referred

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult subjets: Adult subjets diagnosed with bronchiectasis by high-resolution computed tomography with symptomatology in stable phase, matched by by sex and age with healthy subjects.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Pain mechanisms and their clinical impact in patients with bronchiectasis have not been investigated yet. The aim of the research is to assess the presence of central pain mechanisms in patients with bronchiectasis using the Quantitative Sensory Testing (QST) assumptions.

DETAILED DESCRIPTION:
Background and objective:

Recent findings suggest that pain can play an important role in terms of physical activity limitation in respiratory patients. Nevertheless, pain mechanisms and their clinical impact in patients with bronchiectasis have not been investigated yet. The objective of the observational study is to determine the somatosensorial profile in order to assess the presence of central pain mechanisms in patients with bronchiectasis.

Methodology:

Repeated-measures prospective cross-sectional study. A sample of patients diagnosed with bronchiectasis will be recruited and matched by age and sex with healthy controls. Pressure pain thresholds (PPTs), conditioned pain modulation (CPM) and referral pain will be assessed before and after the Incremental Shuttle Walking test (ISW). Levels of physical activity will be assessed using accelerometry during a 7-days period. Sleep quality (Pittsburgh sleep quality test), level of catastrophizing (Pain Catastrophizing Scale), level of sensitization (Central Sensitization Inventory) and level of anxiety and depression (Hospital Anxiety and Depression) will be assessed. The assessments will be done twice: 1) at baseline; and 2) at 6 months follow-up period.

ELIGIBILITY:
Bronchiectasis Group

Inclusion Criteria:

* Diagnosis of bronchiectasis by high-resolution computed tomography.
* Ability to understand and perform all the clinical procedure.
* Acquisition of informed consent.

Exclusion Criteria:

* Diagnosis or clinical suspicion of cystic fibrosis by genetic test or sweat electrolytes test.
* Diagnosis of rheumatic disease.
* Being on a waiting list for lung transplantation.
* Thoraco-abdominal surgery in the last 6 months.
* Chronic use of pain medication.

Control Group

Inclusion Criteria:

* Healthy subjects matched by age and sex with Bronchiectasis Group's subjects

Exclusion Criteria:

* Be taking pain medication.
* Presence of pain condition or pathology.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with bronchiectasis by high-resolution computed tomography with symptomatology in stable phase.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Referred pain area | Baseline
  Amount of pixels painted in an electronic body chart (Navigate Pain, Aalborg, Denmark) after supra threshold pain stimulus (STPS) in infraspinatus muscle.

SECONDARY OUTCOMES:
Number of body areas affected by referred pain | Baseline
  Body chart is divided in 15 regions and the frequency of pain in each one is registered after STPS
Pain intensity after supra threshold pain stimulus (STPS) | Baseline
  Level of pain in a visual analogue scale from 0 to 10 after STPS
Pressure pain thresholds (PPTs) | Baseline
  Level of pressure tolerated by the patient just before feel pain. The pressure is done with an algometer (SB-MEDIC Electronics, Solna, Sweden). PPTS will be assessed bilaterally in infraspinatus, supraspinatus and medial gastrocnemius muscles.
PPTs with a Conditioned Pain Modulation (CPM) pressure stimulus | Baseline
  Level of pressure tolerated by patient just before feel pain. The conditionated pressure stimulus is preform by a blood pressure cuff. CPM will be assessed bilaterally in infraspinatus, supraspinatus and medial gastrocnemius muscles.
Total physical activity time | 7 days period
  Total time spent per day in physical activities at different intensities equal or superior to 100 counts per minute (≥100 cpm), obtained by accelerometry (Actigraph gt3x+).
Sedentary behaviour time | 7 days period
  Total time spent per day in physical activities at different intensities inferior to 100 cpm (<100 cpm).
Light physical activity time | 7 days period
  Total time spent per day in physical activities at intensities between 100 and 1951 cpm (100-1951 cpm).
Moderate-Vigorous physical activity time | 7 days period
  Total time spent per day in physical activities at intensities equal or superior to 1952 cpm (≥1952 cpm).
Level of catastrophizing | Baseline
  Punctuation obtained in Pain Catastrophizing Scale (PCS). It comprises 13 items which focus on thoughts and feelings encountered while experiencing pain. Each item is scored from 0 (not at all) to 4 (all the time) with a total PCS score range from 0-52 points, where higher scores indicating higher levels of pain catastrophizing.
Level of sensitization | Baseline
  Punctuation obtained in Central Sensitization Inventory (CSI). CSI assesses 25 health-related symptoms common to Central Sensitivity Syndromes. Responses are recorded about the frequency of each symptom, with a Likert scale from 0 (never) to 4 (always), resulting in a total possible score of 100. Higher scores are associated with a higher degree of self-reported symptomology.
Level of anxiety and depression | Baseline
  Punctuation obtained in Hospital Anxiety and Depression (HAD). The HAD is a 14-item self-report scale measuring the presence of symptoms of both anxiety (seven items) and depression (seven items) during the past week. Each item is scored from 0 to 3, so the final score for each subscale is between 0 and 21. The majority of the studies use the cutoffs of 7/8 for possible and 10/11 for probable anxiety or depression.
Quality of sleep | Baseline
  Punctuation obtained in Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month in clinical populations. Each sleep component yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. Sleep component scores were summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Level of resilience | Baseline
  Punctuation obtained in Brief Resilience Scale (BRS). This is a 6-item self-report scale with a 5-point response scale ranging from 1 (strongly disagree) to 5 (strongly agree). A higher score indicates a higher degree of resilience.
Distance in ISW test | Baseline
  Meters reached in the ISW test.
Changes in referred pain area | Baseline and after 6 months follow-up
  Amount of pixels painted in an electronic body chart (Navigate Pain, Aalborg, Denmark) after supra threshold pain stimulus (STPS) in infraspinatus muscle.
Changes in number of body areas affected by referred pain | Baseline and after 6 months follow-up
  Body chart is divided in 15 regions and the frequency of pain in each one is registered after STPS
Changes in pain intensity after supra threshold pain stimulus (STPS) | Baseline and after 6 months follow-up
  Level of pain in a visual analogue scale from 0 to 10 after STPS.
Changes in pressure pain thresholds (PPTs) | Baseline and after 6 months follow-up
  Level of pressure tolerated by the patient just before feel pain. The pressure is done with an algometer (SB-MEDIC Electronics, Solna, Sweden)
Changes in Pressure Pain Thresholds (PPTs) with a Conditioned Pain Modulation (CPM) pressure stimulus | Baseline and after 6 months follow-up
  Level of pressure tolerated by patient just before feel pain. The conditionated pressure stimulus is preform by a blood pressure cuff

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad San Jorge, Villanueva de Gállego, Zaragoza, Spain